CLINICAL TRIAL: NCT01334723
Title: Demonstrating the Clinical and Economic Benefit of 5 Alpha Reductase Inhibitor Adherence in Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114482
Record Dates: First submitted 2011-04-07; First posted 2011-04-13 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia, enlarged prostate, 5-alpha-reductase inhibitor, adherence, surgery, acute urinary retention
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — 5-alpha Reductase Inhibitors; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Acute Urinary Retention: This subset of the Integrated Health Care Information Solutions (ICHIS) benign prostate hyperplasia (BPH) study population was used to assess acute urinary retention as a clinical outcome.
  Interventions: Drug: Adherent with 5-alpha-reductase inhibitor (5ARI) therapy; Drug: Non-adherent to 5ARI therapy
- Prostate Surgery: This subset of the ICHIS BPH study population was used to assess surgery as a clinical outcome.
  Interventions: Drug: Adherent with 5-alpha-reductase inhibitor (5ARI) therapy; Drug: Non-adherent to 5ARI therapy

INTERVENTIONS:
Drug: Adherent with 5-alpha-reductase inhibitor (5ARI) therapy — Patient with BPH who are adherent to 5ARI therapy (Adherence will be calculated using a medication possession ratio (MPR); 3 MPR threshold values of 70%, 75%, and 80% will be evaluated.)
  Other Names: Proscar® is a registered trademark of Merck; Avodart® is a registered trademark of GlaxoSmithKline
Drug: Non-adherent to 5ARI therapy — Patients with BPH non-adherent to 5ARI therapy (Adherence will be calculated using a MPR; 3 MPR threshold values of 70%, 75%, and 80% will be evaluated.)
  Other Names: Proscar® is a registered trademark of Merck; Avodart® is a registered trademark of GlaxoSmithKline

SUMMARY:
This retrospective study aims to quantify the relationship between 5-alpha-reductase inhibitor (5ARI) adherence / length of therapy and the likelihood of acute urinary retention (AUR) or prostate surgery in patients with benign prostatic hyperplasia (BPH) as well as the economic impact associated with these medical encounters. The Integrated Health Care Information Solutions (IHCIS) database will be utilized for this study (2000-2006).

ELIGIBILITY:
Inclusion Criteria:

* Male
* aged 50 years or older
* a diagnostic claim of BPH
* prescription claim for a 5ARI for at least 60 days during the observation period.
* continuously eligible for 6 months prior to and at least 6 months after index date.

Exclusion Criteria:

* prostate cancer
* any prostate-related surgical procedure prior to index date

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 50 years or older with a diagnostic claim of BPH and prescription claim for a 5ARI for at least 60 days during the observation period. Patients will be required to be continuously eligible for 6 months prior to and at least 6 months after index date.
Sampling Method: Non-Probability Sample
Enrollment: 35032 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study utilized retrospective claims data from the Integrated Healthcare HealthCare Information Services, Inc. (IHCIS) database, a nationally representative managed care database that represents over 30 healthplans and more than 25 million lives.
Pre-assignment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Acute Urinary Retention Outcomes Cohort: This subset of the Integrated Health Care Information Solutions (ICHIS) benign prostate hyperplasia (BPH) study population was used to assess acute urinary retention as a clinical outcome.
- Prostate Surgery Outcomes Cohort: This subset of the ICHIS BPH study population was used to assess surgery as a clinical outcome.
Period: Overall Study
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Started | 17293 | 17739
Completed | 17293 | 17739
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort | Total
Number analyzed (Participants) | 17293 | 17739 | 35032
Age, Customized [Number; unit: participants]
  Age >= 50 | 17293 | 17739 | 35032
  Age < 50 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17293 | 17739 | 35032

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Risk of Acute Urinary Retention and Surgery Based on an MPR Threshold of 70%
Description: Claims-based definition of acute urinary retention (AUR) and surgery based on the presence of an ICD-9-CM code of 599.6x, 788.20, or 788.29 and CPT procedure codes, respectively. For this analysis, we evaluated the association between compliance with 5-ARI therapy (measured by medication possession ratio [MPR]) and risk of AUR or surgery. MPR was calculated as the number of days that 5-ARI therapy was taken divided by the total number of follow-up days. For this analysis, the threshold for compliance was set at MPR = 70%.
Time Frame: The 5 and a half year period from January 1, 2000 to June 30, 2006
Population: Enrolled Population: participants in the IHCIS database with a diagnosis of benign prostate hyperplasia or enlarged prostate as indicated by ICD-9-CM code on claims (222.2x or 600.xx). Participants were included if they had at least 60 days of 5-ARI therapy during the enrollment period, 6 months of continuous enrollment, and no prior surgery.
Measure: Number; unit: participants
Groups:
- Acute Urinary Retention Outcomes Cohort, MPR <=70%: Participants in the acute urinary retention outcomes cohort with an MPR <=70%
- Acute Urinary Retention Outcomes Cohort, MPR >70%: Participants in the acute urinary retention outcomes cohort with an MPR >70%
- Prostate Surgery Outcomes Cohort, MPR <=70%: Participants in the prostate surgery outcomes cohort with an MPR <=70%
- Prostate Surgery Outocomes Cohort, MPR >70%: Participants in the prostate surgery outcomes cohort with an MPR >70%
Arm/Group | Acute Urinary Retention Outcomes Cohort, MPR <=70% | Acute Urinary Retention Outcomes Cohort, MPR >70% | Prostate Surgery Outcomes Cohort, MPR <=70% | Prostate Surgery Outocomes Cohort, MPR >70%
Number analyzed (Participants) | 7651 | 9642 | 7386 | 10353
participants
  Number of Participants with AUR and Surgery | 2140 | 1587 | 481 | 331
  Number of Participants without AUR and Surgery | 5511 | 8055 | 6905 | 10022
Statistical Analysis 1: Comparison: Acute Urinary Retention Outcomes Cohort, MPR <=70% vs Acute Urinary Retention Outcomes Cohort, MPR >70%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.380, 95% CI [0.350 to 0.412] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery
Statistical Analysis 2: Comparison: Prostate Surgery Outcomes Cohort, MPR <=70% vs Prostate Surgery Outocomes Cohort, MPR >70%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.294, 95% CI [0.235 to 0.368] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery

2. Primary Outcome: Number of Participants With Risk of Acute Urinary Retention and Surgery Based on an MPR Threshold of 75%
Description: Claims-based definition of AUR and surgery based on the presence of an ICD-9-CM code of 599.6x, 788.20, or 788.29 and CPT procedure codes, respectively. For this analysis, we evaluated the association between compliance with 5-ARI therapy (measured by medication possession ratio [MPR]) and risk of AUR and surgery. MPR was calculated as the number of days that 5-ARI therapy was taken divided by the total number of follow-up days. For this analysis, the threshold for compliance was set at MPR = 75%.
Time Frame: Up to one year following the first pharmacy claim for 5ARI therapy or medical encounter for AUR or prostate surgery in the 5 and a half year period from January 1, 2000 to June 30, 2006
Population: Enrolled Population
Measure: Number; unit: participants
Groups:
- Acute Urinary Retention Outcomes Cohort, MPR <=75%: Among the Participants in the acute urinary retention outcomes cohort with an MPR <=75%
- Acute Urinary Retention Outcomes Cohort, MPR >75%: Participants in the acute urinary retention outcomes cohort with an MPR >75%
- Prostate Surgery Outcomes Cohort, MPR <=75%: Participants in the prostate surgery outcomes cohort with an MPR <=75%
- Prostate Surgery Outcomes Cohort, MPR >75%: Participants in the prostate surgery outcomes cohort with an MPR >75%
Arm/Group | Acute Urinary Retention Outcomes Cohort, MPR <=75% | Acute Urinary Retention Outcomes Cohort, MPR >75% | Prostate Surgery Outcomes Cohort, MPR <=75% | Prostate Surgery Outcomes Cohort, MPR >75%
Number analyzed (Participants) | 10413 | 6880 | 11107 | 6632
participants
  Number of Participants with AUR and surgery | 2755 | 1277 | 627 | 185
  Number of Participants without AUR and surgery | 7658 | 5603 | 10480 | 6447
Statistical Analysis 1: Comparison: Acute Urinary Retention Outcomes Cohort, MPR <=75% vs Acute Urinary Retention Outcomes Cohort, MPR >75%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.613, 95% CI [0.562 to 0.668] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery
Statistical Analysis 2: Comparison: Prostate Surgery Outcomes Cohort, MPR <=75% vs Prostate Surgery Outcomes Cohort, MPR >75%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.542, 95% CI [0.427 to 0.689] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery

3. Primary Outcome: Number of Participants With Risk of Acute Urinary Retention and Surgery Based on an MPR Threshold of 80%
Description: Claims-based definition of AUR and surgery based on the presence of an ICD-9-CM code of 599.6x, 788.20, or 788.29 and CPT procedure codes, respectively. For this analysis, we evaluated the association between compliance with 5-ARI therapy (measured by medication possession ratio [MPR]) and risk of AUR and surgery. MPR was calculated as the number of days that 5-ARI therapy was taken divided by the total number of follow-up days. For this analysis, the threshold for compliance was set at MPR = 80%.
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Number; unit: participants
Groups:
- Acute Urinary Retention Outcomes Cohort, MPR <=80%: Participants in the acute urinary retention outcomes cohort with an MPR <=80%
- Acute Urinary Retention Outcomes Cohort, MPR >80%: Participants in the acute urinary retention outcomes cohort with an >80%
- Prostate Surgery Outcomes Cohort, MPR <=80%: Participants in the prostate surgery outcomes cohort with an MPR <=80%
- Prostate Surgery Outcomes Cohort, MPR >80%: Participants in the prostate surgery outcomes cohort with an MPR >80%
Arm/Group | Acute Urinary Retention Outcomes Cohort, MPR <=80% | Acute Urinary Retention Outcomes Cohort, MPR >80% | Prostate Surgery Outcomes Cohort, MPR <=80% | Prostate Surgery Outcomes Cohort, MPR >80%
Number analyzed (Participants) | 11787 | 5506 | 11953 | 5786
participants
  Number of Participants with AUR and surgery | 2812 | 915 | 627 | 185
  Number of Participants without AUR and surgery | 8975 | 4591 | 11326 | 5601
Statistical Analysis 1: Comparison: Acute Urinary Retention Outcomes Cohort, MPR <=80% vs Acute Urinary Retention Outcomes Cohort, MPR >80%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.519, 95% CI [0.472 to 0.570] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery
Statistical Analysis 2: Comparison: Prostate Surgery Outcomes Cohort, MPR <=80% vs Prostate Surgery Outcomes Cohort, MPR >80%; Test type: Superiority or Other; Hazard Ratio (HR) = 0.436, 95% CI [0.333 to 0.570] — A time-to-event analysis was used to evaluate the likelihood of AUR or prostate surgery

4. Secondary Outcome: Mean Length of 5-ARI Therapy
Description: In this analysis, we evaluated the association between 5-ARI length of therapy and risk of acute urinary retention and prostate surgery.
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Number analyzed (Participants) | 17293 | 17739
days | 276.8 (89.1) | 289.5 (85.1)

5. Secondary Outcome: Mean BPH-Related Costs for Participants With an MPR >=70% Versus <70%
Description: In this analysis, we evaluated mean BPH-related costs per month for participants with an MPR of >=70% versus <70%. Mean costs were evaluated by month on therapy for BPH-related medical costs (defined as any claim with a primary ICD-9-CM code of 222.2 or 600.xx).
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars per month
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Number analyzed (Participants) | 17293 | 17739
United States dollars per month
  MPR >=70% | 23.56 (10.45) | 24.40 (10.64)
  MPR <70% | 35.25 (15.64) | 38.59 (16.83)

6. Secondary Outcome: Mean BPH-Related Costs for Participants With an MPR >=75% Versus <75%
Description: In this analysis, we evaluated mean BPH-related costs per month for participants with an MPR of >=75% versus <75%. Mean costs were evaluated by month on therapy for BPH-related medical costs (defined as any claim with a primary ICD-9-CM code of 222.2 or 600.xx).
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars per month
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Number analyzed (Participants) | 17293 | 17739
United States dollars per month
  MPR >=75% | 27.12 (12.05) | 27.14 (12.11)
  MPR <75% | 29.64 (13.17) | 32.37 (14.44)

7. Secondary Outcome: Mean BPH-Related Costs for Participants With an MPR >=80% Versus <80%
Description: In this analysis, we evaluated mean BPH-related costs per month for participants with an MPR of >=80% versus <80%. Mean costs were evaluated by month on therapy for BPH-related medical costs (defined as any claim with a primary ICD-9-CM code of 222.2 or 600.xx).
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars per month
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Number analyzed (Participants) | 17293 | 17739
United States dollars per month
  MPR >=80% | 24.24 (10.8) | 23.02 (10.19)
  MPR <80% | 30.83 (13.73) | 33.95 (15.03)

8. Secondary Outcome: BPH-Related Costs for Every 30 Days of 5-ARI Therapy
Description: In this analysis, we evaluated mean BPH-related costs for every 30 days of 5-ARI therapy. Mean costs were evaluated by month on therapy for BPH-related medical costs (defined as any claim with a primary ICD-9-CM code of 222.2 or 600.xx).
Time Frame: as for outcome 2
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: United States dollars per month
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Number analyzed (Participants) | 17293 | 17739
United States dollars per month | 28.08 (145.40) | 29.89 (156.22)

ADVERSE EVENTS:
Description: This was a retrospective database study, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | Acute Urinary Retention Outcomes Cohort | Prostate Surgery Outcomes Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.